CLINICAL TRIAL: NCT05304182
Title: Clinical Study - ES 900 - 2020-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Haag-Streit AG (Industry)
Collaborators: Aravind Eye Hospitals, India (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 1023703
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Cataract
Keywords: Optical Biometry; Corneal Topography
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: There are two identical arms in this study: pre-operative and post-operative. Every participant starts in the pre-operative arm and crosses over to the post-operative arm. During both arms, each study subject undergoes the experimental intervention and the control intervention.
  The study objective is to assess the clinical performance of the investigational device. This assessment is performed by a statistical analysis of the measurement results from the experimental intervention and the control intervention. The surgery is not a study intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Op (Experimental): The experimental intervention is non-invasive optical imaging, in particular digital photography and optical coherence tomography, conducted with the investigational and comparator device, for the purpose of measuring dimensions of the eye.
  Interventions: Device: EYESTAR 900; Device: LENSTAR LS 900
- Post-Op (Active Comparator): The experimental intervention is non-invasive optical imaging, in particular digital photography and optical coherence tomography, conducted with the investigational and comparator device, for the purpose of measuring dimensions of the eye.
  Interventions: Device: EYESTAR 900; Device: LENSTAR LS 900

INTERVENTIONS:
Device: EYESTAR 900 — The EYESTAR 900 is a device developed by Haag-Streit which utilises 3D OCT for quantitative measurements of the geometry of the entire eye, including ocular biometry and corneal topography. It is the most recent in a series of successful biometry devices by Haag-Streit (HS Pachymeter, Lenstar LS 900, LS 900 T-cone and LS 900 APS) and also allows for advanced corneal tomography examinations.
  Other Names: Optical Biometer
Device: LENSTAR LS 900 — The LENSTAR LS 900 is a non-contact device for measurement of biometrical parameters of the eye, aimed to assist the calculation of intraocular lenses (IOLs) prior to intraocular lens implantation. The most common application is in preparation of cataract surgery.
  This device uses OLCR (optical low-coherence reflectometry), an interferometric method to measure intraocular axial distances. Furthermore, it uses digital photography of the anterior section of the eye to measure pupil size and location, as well as the white-to-white distance of the eye. The same photographic unit, in conjunction with a specific illumination pattern, is used to measure the corneal curvature - this measurement is known as 'keratometry', or, more specifically, 'automated keratometry'.
  Other Names: Optical Biometer

SUMMARY:
EYESTAR 900 is a device developed by Haag-Streit which utilises 3D OCT for quantitative measurements of the geometry of the entire eye, including ocular biometry and corneal topography. It is the most recent in a series of successful biometry devices by Haag-Streit (HS Pachymeter, Lenstar LS 900, LS 900 T-cone and LS 900 APS) and also allows for advanced corneal tomography examinations. The EYESTAR 900 is CE marked.

These measurement results of this device are used for the planning of the medical treatment of patients. Depending on the application, the benefits of this device may include improved visual acuity (after cataract surgery), reduced risk of complications (after refractive surgery or implant of a phakic intraocular lens), early identification of pathological deformations of the cornea (keratoconus detection).

The primary objective of this clinical trial is to assess the clinical performance of the investigational device in dense cataracts. To that end, for each measurand, the in-vivo repeatability will be quantified, as well as limits of agreement and the mean measurement deviation, with respect to the current gold standard device.

As a secondary objective of the study, raw measurement data will be collected to allow for the improvement of existing algorithms, development of additional measurands and for retrospective analysis.

No diseases are studied.

DETAILED DESCRIPTION:
The EYESTAR 900 is a non-contact device for measuring the human eye, consisting of a swept source OCT sub-unit (OCT: optical coherence tomography, a measurement method to acquire tomographic images by optical interferometry) and an imaging system sub-unit.

The OCT sub-unit performs a three-dimensional measurement of all refractive ocular structures in the anterior eye segment (curvatures and locations of the anterior corneal surface, posterior corneal surface, the anterior crystalline lens surface, posterior crystalline lens surface), as well as a one-dimensional measurement of axial eye length. It also generates cross-sectional images of the anterior eye section and the central retina. The measurement is implemented by scanning the eye with a low-power near-infrared laser beam and measuring the light which is back-reflected to the device.

The imaging system sub-unit is used to obtain photographic images of the eye. Based on these images, the keratometry (anterior corneal curvature of the steepest and flattest meridian), the white-to-white distance and the pupil diameter are measured. Additionally, these images can serve to document the locations of special landmarks on the eye, such as blood vessels. The imaging system sub-unit is based on conventional digital photography technology. Illumination for imaging is provided by infrared and white-light LEDs (light emitting diodes). Measurement of keratometry additionally requires measuring the distance to the eye using the OCT sub-unit.

The EYESTAR 900 is designed as standalone-device with integrated PC (personal computer) and display for device operation, measurement acquisition and processing, and presentation of the measurement results. After a patient is placed in front of the device and the chin rest is adjusted, the device can perform the remaining positioning procedures and acquire the measurements in a fully automated manner. Position information is derived from the OCT and digital camera system sub-units.

Both implemented measuring methods, optical coherence tomography (OCT), as well as digital photography are non-invasive, contactless methods. OCT uses a laser beam of λ=1060nm central wavelength and less than 2 mW optical power, which is focussed to a beam diameter of approximately 80µm at the anterior lens plane, and is continuously scanned in the lateral direction. Digital photography uses diffuse illumination of the eye by white-light LEDs (425nm ≤ λ ≤ 725nm) and infrared LEDs with central wavelength λ=850nm. All light sources emit levels that comply with ISO 15004-2 ("Ophthalmic Instruments - Fundamental requirements and test methods - Part 2: Light hazard protection"), under normal operating conditions as well as in case of a single fault condition.

The main application of this device is to acquire biometric measurements of cataractous eyes which are used to calculate suitable intraocular lens power and dimension.

The patient population must be capable of sitting up straight and keeping their head still and their eyes opened. They must be physically and mentally able to cooperate and mentally capable of following the examination. Patients must be at least 18 years old.

The target device user is an ophthalmologist or a trained specialist.

The investigational device EYESTAR 900 is developed and manufactured by HAAG-STREIT AG, Koeniz (Switzerland).

For the duration of the examination (approximately 1-2 minutes), the patient is in contact with the device at following applied parts:

1. the chin rest shell (Edistir RK451 G naturally coated with HAERATEX Aqua 2K-structural coater BW89 10K RAL 9005);
2. the forehead rest band (Saxamid 126-N001 uncoated PA6 white FK 6659 PA);
3. (depending on the subject's requirements) the patient handles (aluminium EN AW-6060 (AlMgSi 0.5) colourless anodized class 20 with sealing chemically polished and sandblasted).

No other contact with body tissues or fluids takes place. No critical biocompatibility issues were identified.

ELIGIBILITY:
Inclusion Criteria:

* voluntary participation
* informed consent
* 35 years of age or older

Exclusion Criteria:

* ineligibility for cataract surgery for any reason, e.g., aphakia
* Disqualifying pathologies:

  * keratoconus
  * corneal astigmatism of more than 3.5 D
  * history of recurrent inflammation or infection of the eye
* Disqualifying corneal conditions:

  * comorbidities,
  * deformations,
  * lesions, or
  * scarring of the cornea
  * acute inflammation or infection of the eye
* Disqualifying treatments:

  * previous refractive surgeries, including PRK and LASIK
  * previous corneal surgeries
  * previous corneal transplants
  * previous intraocular surgeries
* Disqualifying outcomes:

  * failed IOL implantation into the capsular bag

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Dense Cataract Performance | 18 months
  The primary outcome is the performance of the EYESTAR 900 in dense cataracts. Specifically, the highest grade of cataract at which complete measurements can reliably be performed and, consequently, the number of patients measured successfully.

SECONDARY OUTCOMES:
Keratometry | 18 months
  The limits of agreement and the confidence interval of difference in comparison with the LENSTAR 900.
Axial Length | 18 months
  The limits of agreement and the confidence interval of difference in comparison with the LENSTAR 900.
White-to-White Imaging | 18 months
  The limits of agreement and the confidence interval of difference in comparison with the LENSTAR 900.
Anterior Corneal Elevation | 18 months
  The limits of agreement and the confidence interval of difference in comparison with the LENSTAR 900.
Anterior Corneal Axial Curvature | 18 months
  The limits of agreement and the confidence interval of difference in comparison with the LENSTAR 900.
Anterior Corneal Tangential Curvature | 18 months
  The limits of agreement and the confidence interval of difference in comparison with the LENSTAR 900.
Posterior Corneal Elevation | 18 months
  The limits of agreement and the confidence interval of difference in comparison with the LENSTAR 900.
Posterior Corneal Axial Curvature | 18 months
  The limits of agreement and the confidence interval of difference in comparison with the LENSTAR 900.
Posterior Corneal Tangential Curvature | 18 months
  The limits of agreement and the confidence interval of difference in comparison with the LENSTAR 900.
Corneal Pachymetry | 18 months
  The limits of agreement and the confidence interval of difference in comparison with the LENSTAR 900.
Simulated Anterior Keratometry | 18 months
  The limits of agreement and the confidence interval of difference in comparison with the LENSTAR 900.
Simulated Posterior Keratometry | 18 months
  The limits of agreement and the confidence interval of difference in comparison with the LENSTAR 900.

CONTACTS AND LOCATIONS:
Overall Officials: Haripriya Aravind, MD, Principal Investigator — Aravind Eye Hospitals; Thomas Beutler, Dipl. Ing., Study Director — Haag-Streit AG; Julian Kool van Langenberghe, ing., Study Chair — Haag-Streit AG
Locations (1):
- Aravind Eye Hospitals, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No